CLINICAL TRIAL: NCT00850434
Title: Study of an Improved Automatic CPAP Algorithm for the Treatment of Obstructive Sleep Apnea
Brief Title: Improved Automatic CPAP Algorithm to Treat Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MA20041125
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- modified autoset (Experimental): the modified AutoSet responds to different breathing patterns than the standard AutoSet, to treat OSA. Participants in this arm will trial the modified AutoSet for one night, and the standard AutoSet for one night, in a randomised order
  Interventions: Device: Modified AutoSet Algorithm; Device: Standard AutoSet Algorithm
- standard AutoSet (Active Comparator): The standard autoset treat OSA by using pressure increases to overcome abnormal breathing patterns. Patients in this arm will use the standard AutoSet for one night and the modified AutoSet for one night, in a randomised order
  Interventions: Device: Modified AutoSet Algorithm; Device: Standard AutoSet Algorithm

INTERVENTIONS:
Device: Modified AutoSet Algorithm — The modified AutoSet algorithm responds to more patient "non-normal" flow types than the standard AutoSet algorithm
  Other Names: Enhanced AutoSet algorithm
Device: Standard AutoSet Algorithm — The standard AutoSet used for treatment of OSA

SUMMARY:
The purpose of this study is to compare a modified AutoSet algorithm running on research hardware versus the traditional AutoSet algorithm running on an S7 AutoSet Spirit. The study will determine if the modified AutoSet algorithm reacts appropriately to obstructive apnoeas and hypopnoeas and provides suitable levels of positive airway pressure compared to the S7 AutoSet Spirit.

The hypothesis is that the modified AutoSet algorithm will be more efficacious than the traditional AutoSet algorithm

DETAILED DESCRIPTION:
Subjects in the trial will spend 2 nights in a sleep laboratory being monitored with a full montage polysomnograph (PSG) with each of the algorithms providing positive airway pressure therapy. The PSG records EEG, EMG, EOG, patient airflow, respiratory effort, blood oxygen saturation, and body position.

In a randomised order each subject will spend one night being treated by the modified AutoSet algorithm and a second night being treated by the traditional AutoSet algorithm.

The subjects will be blinded to which therapy they are receiving and the scorer of the PSG will also be blinded to which therapy is being used.

ELIGIBILITY:
Inclusion Criteria:

* PSG-confirmed diagnosis of OSA, showing an apnoea-hypopnoea index (AHI) of at least 15 events/hr and an obstructive apnoea index (OAI) of at least 5 events/hr.
* On CPAP therapy (fixed pressure or autoCPAP) for at least 1 month.
* Using a ResMed mask (this requirement applies only to phase 2 of the trial) without significant discomfort for at least 2 weeks.
* Age between 18 and 70 years.
* Written informed consent.

Exclusion Criteria:

* Unstable medical condition, including unstable angina, myocardial infarction within previous 6 months, cardiac failure NYHA grades III and IV, epilepsy, psychiatric disturbance.
* Respiratory insufficiency, defined as arterial CO2 greater than 50 mm Hg during the daytime or arterial oxygen saturation less than 90% when asleep and breathing room air on effective CPAP therapy.
* Recent severe epistaxis.
* History of spontaneous pneumothorax.
* History of regurgitation of gastric contents during sleep.
* Unable to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Physiological sleep signals including EEG, Sp02, respiratory effort and nasal flow, will be recorded, analysed and reported in the form of a series of indices, which are the outcome variables of the study. | Two consecutive nights
  sleep signals taken from overnight polysomnography recordings

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed / University of NSW
Locations (1):
- Sleep & Chest Disorders Centre, Sydney, New South Wales, Australia